CLINICAL TRIAL: NCT03753490
Title: ABC-Risk Scores for Reduction of Stroke and Mortality in Atrial Fibrillation - a Multicenter, Registry-based, Randomized Controlled Parallel-group Open-label Study
Brief Title: ABC-Scores for Reduction of Stroke and Mortality in Atrial Fibrillation - The ABC-AF Study
Acronym: ABC-AF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Swedish Foundation for Strategic Research (Other); Swedish Heart Lung Foundation (Other); Roche Diagnostics GmbH (Industry); The Swedish Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1011455
Record Dates: First submitted 2018-11-08; First posted 2018-11-27 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ABC score guided therapy (Other): Individual treatment recommendations based on the ABC-scores for stroke and bleeding.
  Interventions: Other: ABC score guided therapy
- Standard care (Other): Management according to local practice, national and international guidelines.
  Interventions: Other: Standard care

INTERVENTIONS:
Other: ABC score guided therapy — In the ABC arm, individual treatment recommendations based on the ABC-scores for stroke and bleeding including non-vitamin K oral anticoagulant or no anticoagulant treatment, and other drugs and interventions, to improve stroke free survival.
  Arms: ABC score guided therapy
Other: Standard care — In the standard care arm, management according to local practice, national and international guidelines, including the potential use of traditional clinical risk scores for stroke and/or bleeding, anticoagulant treatment and other treatments and interventions.
  Arms: Standard care

SUMMARY:
The primary study objective is to evaluate if personalized treatment by decision support, based on the biomarker-based risk prediction (ABC-scores) guided strategy, reduces the occurrence of the composite outcome of stroke or death in patients with atrial fibrillation. Approximately 6500 patients will be randomized 1:1 to ABC risk score guided therapy or standard care.

ELIGIBILITY:
Inclusion criteria:

1. Patients with diagnosis of atrial fibrillation, including newly diagnosed, with or without current oral anticoagulant treatment
2. Signed informed consent

Exclusion criteria:

1. Contraindication for any oral anticoagulant, according to the SmPC (in Sweden FASS)
2. Indication for oral anticoagulant treatment beyond atrial fibrillation, e.g. venous thromboembolism and/or mechanical heart valve prosthesis
3. Currently on treatment with a non-vitamin K antagonist oral anticoagulant (NOAC) and not eligible for change of NOAC drug e.g. drug-drug interactions
4. Concomitant dual antiplatelet treatment
5. Acute coronary syndrome (myocardial infarction or unstable angina) within the last 30 days
6. Participation in anti-thrombotic pharmaceutical trial
7. Planned for AF ablation or AF surgery
8. Haemoglobin <90 g/L
9. Patients who, in the opinion of the investigator, cannot or will not comply with the requirements of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3933 (Estimated)
Dates: Start 2018-10-25 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Composite of Stroke or Death | From the date of enrolment through study completion, minimum follow-up 2 years.

SECONDARY OUTCOMES:
Major Bleeding | From the date of enrolment through study completion, minimum follow-up 2 years.
Stroke | From the date of enrolment through study completion, minimum follow-up 2 years.
Death | From the date of enrolment through study completion, minimum follow-up 2 years.
Myocardial Infarction | From the date of enrolment through study completion, minimum follow-up 2 years.
Heart Failure | From the date of enrolment through study completion, minimum follow-up 2 years.
Health Economics | From the date of enrolment through study completion, minimum follow-up 2 years.
  Mean differences in health care cost, and 2-year quality-adjusted survival based on EuroQol-5D-5L between the treatment groups, combined into an incremental cost-effectiveness ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Oldgren, MD, PhD, Study Director — Uppsala Clinical Reseach Center, UCR
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oldgren J, Hijazi Z, Arheden H, Bjorkenheim A, Frykman V, Janzon M, Ravn-Fischer A, Renlund H, Sjalander A, Akerfeldt T, Wallentin L. Biomarker-Based ABC-AF Risk Scores for Personalized Treatment to Reduce Stroke or Death in Atrial Fibrillation: A Registry-Based, Multicenter, Randomized, Controlled Study. Circulation. 2025 Nov 25;152(21):1457-1469. doi: 10.1161/CIRCULATIONAHA.125.076725. Epub 2025 Aug 30. PMID 40884774